CLINICAL TRIAL: NCT06989983
Title: An Open-Label, Two-Period Study Designed to Assess the Mass Balance Recovery, Absorption, Metabolism, Excretion of [14C]AZD5462 and the Absolute Bioavailability of AZD5462 in Healthy Male Participants
Brief Title: A Study Designed to Assess the Mass Balance Recovery, Absorption, Metabolism, Excretion of [14C]AZD5462 and the Absolute Bioavailability of AZD5462
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9090C00009
Record Dates: First submitted 2025-05-05; First posted 2025-05-25 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD5462 (Experimental): In Period 1, participants will receive one oral dose of [14C]AZD5462.
  In Period 2, participants will receive one oral dose of AZD5462 and one intravenous dose of [14C]AZD5462.
  Interventions: Drug: AZD5462 film-coated tablet; Drug: [14C]AZD5462 Solution for Infusion; Drug: [14C]AZD5462 Oral Solution

INTERVENTIONS:
Drug: AZD5462 film-coated tablet — Oral, fasted
  Other Names: AZD5462
Drug: [14C]AZD5462 Solution for Infusion — Intravenous, fasted
  Other Names: AZD5462
Drug: [14C]AZD5462 Oral Solution — Oral, fasted
  Other Names: AZD5462

SUMMARY:
A study to investigate how the body breaks down and gets rid of the test medicine, AZD5462.

To help investigate this, the test medicine is radiolabelled, which means that the test medicine has a radioactive component (carbon-14), which helps us to track where the test medicine is in the body. The safety and tolerability of the test medicine will also be studied.

DETAILED DESCRIPTION:
This is an open-label, two-period study designed to assess the mass balance recovery, absorption, metabolism, excretion of [14C]AZD5462 and the absolute bioavailability of AZD5462 in healthy male participants.

The study will take place at 1 site in Nottingham, and enrol 8 healthy men aged 30-65 years. The study will include 2 Periods:

* In Period 1 volunteers will receive a single dose of radiolabelled test medicine as a liquid by mouth.
* In Period 2 volunteers will receive a single dose of the test medicine as capsules by mouth and shortly afterwards, a very tiny dose of radiolabelled study medicine by injection into a vein.

The participants will be resident in the clinical unit throughout both study periods for a total of 12 nights. The total study duration is approximately up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 30 to 65 years inclusive
* BMI in the range 18.0 - 32.0 kg/m2 inclusive and body weight ≥ 50 kg and ≤ 100 kg
* Regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History or presence of clinically significant gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity
* History of active malignancy within 2 years, or under investigation for any form of cancer
* Participants who do not have suitable veins for multiple venepunctures/cannulation
* Clinically significant abnormal clinical chemistry, haematology or urinalysis
* Any clinically significant abnormalities in vital signs
* Any clinically significant abnormalities on 12-lead ECG
* Abnormal renal function
* Radiation exposure exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years, occupationally exposed worker, or have been administered IMP in a radiolabelled ADME study in the last 12 months.
* Use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals
* Current smokers or known or suspected history of alcohol or drug abuse
* Excessive intake of caffeine-containing drinks or food

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Amount of AZD5462 excreted (Ae) - Period 1 | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Mass balance recovery of total radioactivity of [14C]AZD5462 in urine and faecal samples
Amount of AZD5462 excreted expressed as a percentage of the dose administered (Fe) - Period 1 | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Mass balance recovery of total radioactivity of [14C]AZD5462 in urine and faecal samples
Cumulative amount of AZD5462 excreted (CumAe) - Period 1 | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Mass balance recovery of total radioactivity of [14C]AZD5462 in urine and faecal samples
Cumulative amount of AZD5462 excreted expressed as a percentage of the dose administered (CumFe) - Period 1 | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Mass balance recovery of total radioactivity of [14C]AZD5462 in urine and faecal samples
Absolute bioavailability - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  Absolute bioavailability (F) based on AUC0-inf of oral and IV administration, adjusted for dose

SECONDARY OUTCOMES:
Time of maximum observed concentration (tmax) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Maximum observed concentration (Cmax) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Area under the curve from time 0 to the time of last measurable concentration (AUC0-t) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUC0-extrap) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Terminal elimination half-life (t1/2) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
First order rate constant associated with the terminal (log-linear) portion of the curve (λz) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown (CL/F) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Renal clearance calculated using plasma AUC (CLR) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma and urine
Apparent volume of distribution based on the terminal phase calculated using AUC(0 inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown (Vz/F) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma and urine
Area under the curve (AUC) of circulating plasma total radioactivity (TR) or accounting for 10% or more of the dose in excreta - Period 1 | Plasma, urine and faecal samples from pre-dose until 168 hours post-dose
  Identification of the chemical structure of each metabolite accounting for more than 10% by AUC of circulating TR or accounting for 10% or more of the dose in urine and faeces
Blood:plasma concentration ratios - Period 1 | Whole blood samples and plasma samples collected from pre-dose until 168 hours post-dose
  Blood:plasma concentration ratios of total radioactivity
Amount of unchanged AZD5462 excreted in urine (Ae) - Period 2 | Urine sample collection from pre-dose to 72 hours post-dose
  Recovery of total radioactivity of [14C]AZD5462 in urine
Amount of unchanged AZD5462 excreted in urine expressed as a percentage of the radioactive dose administered (Fe) - Period 2 | Urine sample collection from pre-dose to 72 hours post-dose
  Recovery of total radioactivity of [14C]AZD5462 in urine
Cumulative amount of unchanged AZD5462 excreted in urine (CumAe) - Period 2 | Urine sample collection from pre-dose to 72 hours post-dose
  Recovery of total radioactivity of [14C]AZD5462 in urine
Cumulative amount of unchanged AZD5462 excreted in urine expressed as a percentage of the radioactive dose administered (CumFe) - Period 2 | Urine sample collection from pre-dose to 72 hours post-dose
  Recovery of total radioactivity of [14C]AZD5462 in urine
Area under the curve from time 0 extrapolated to infinity (AUC0-inf) for AZD5462 and total radioactivity - Period 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Time of maximum observed concentration (tmax) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Maximum observed concentration (Cmax) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Area under the curve from time 0 extrapolated to infinity (AUC0-inf) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Area under the curve from time 0 to the time of last measurable concentration (AUC0-t) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUC0-extrap) for AZD5462 and [14C]AZD5462- Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Terminal elimination half-life (t1/2) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
First order rate constant associated with the terminal (log-linear) portion of the curve (λz) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Total body clearance calculated after a single IV administration (CL) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown (CL/F) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single IV administration (Vz) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Apparent volume of distribution at steady state after a single IV administration (Vss) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Apparent volume of distribution based on the terminal phase calculated using AUC(0 inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown (Vz/F) for AZD5462 and [14C]AZD5462 - Period 2 | Plasma sample collection from pre-dose to 72 hours post-dose
  PK of AZD5462 and [14C]AZD5462 in plasma
Number of subjects with treatment-related adverse events - Periods 1 and 2 | Through study duration, an average of 7 weeks
  To provide additional safety and tolerability information for AZD5462

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MBChB, MRCS (Ed), Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual participant-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/